CLINICAL TRIAL: NCT03514108
Title: A Randomized, Double-blind, Placebo Controlled Study (DANHEART): Hydralazine-ISDN in Patients With Chronic Heart Failure - Hydralazine Heart Failure Trial (H-HeFT) and Metformin in Patients With Chronic Heart Failure and Diabetes or Insulin Resistance - Metformin Heart Failure Trial (Met-HeFT)
Brief Title: DANHEART (H-HeFT and Met-HeFT)
Acronym: DANHEART
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Henrik Wiggers (Other)
Collaborators: Danish Heart Foundation (Other); Danish Council for Independent Research (Other); The Danish Regions: Foundation for Medical Research (Unknown); The Novo Nordisk Foundation (Unknown); The Aase og Ejnar Danielsen Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Henrik Wiggers, Professor, Consultant, MD, PhD, DMSc, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DANHEART; 2015-002150-12 (EudraCT Number)
Record Dates: First submitted 2018-02-20; First posted 2018-05-02 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure; Diabetes
Keywords: Heart failure; Diabetes; Insulin resistance; Metformin; Hydralazine; Isosorbide Dinitrate
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus; Insulin Resistance | interventions — isosorbide-hydralazine combination; Metformin

STUDY DESIGN:
Intervention Model Description: Patients can be allocated to either
  1. both Hydralazine Isosorbide Dinitrate / Placebo and Metformin hydrochloride / Placebo
  2. to only Hydralazine Isosorbide Dinitrate / Placebo.
  3. to only Metformin hydrochloride / Placebo.
  Patient characteristics are entered in an electronic CRF. According to in- and exclusion criteria they are randomized in three blocks:
  1. Patients receiving both Hydralazine Isosorbide Dinitrate / Placebo and Metformin hydrochloride / Placebo
  2. Patients receiving only Hydralazine Isosorbide Dinitrate / Placebo and
  3. Patients receiving only Metformin hydrochloride / Placebo
  Analysis will be performed in:
  1. all patients who have received Hydralazine Isosorbide Dinitrate / Placebo (H-HeFT) and
  2. all patients who have received Metformin hydrochloride / Placebo (Met-HeFT)
  The study is event driven. Anticipated: both H-HeFT and Met-HeFT 900, only H-HeFT 400, only Met-HeFT 200 patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Hydralazine Isosorbide Dinitrate (Active Comparator): Tablet BiDil (Hydralazine 37.5 mg/ isosorbide dinitrate (ISDN) 20 mg) 2 tablets x 3 daily.
  Average treatment period 4 years.
  Interventions: Drug: Hydralazine Isosorbide Dinitrate
- Placebo (Hydralazine Isosorbide Dinitrate) (Placebo Comparator): Tablet Placebo 2 tablets x 3 daily. Average treatment period 4 years.
  Interventions: Drug: Placebo Oral Tablet
- Metformin (Active Comparator): Tablet Metformin hydrochloride 500 mg 2 tablets x 2 daily (eGFR 35-60 ml/min: 500 mg x 2 daily). Average treatment period 4 years.
  Interventions: Drug: Metformin Hydrochloride
- Placebo (Metformin) (Placebo Comparator): Tablet Placebo 500 mg 2 tablets x 2 daily (eGFR 35-60 ml/min: 500 mg x 2 daily). Average treatment period 4 years.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Hydralazine Isosorbide Dinitrate — Tablet BiDil (Hydralazine 37.5 mg/ Isosorbide Dinitrate (ISDN) 20 mg) 2 tablets x 3 daily
  Other Names: BiDil
  Arms: Hydralazine Isosorbide Dinitrate
Drug: Placebo Oral Tablet — 2 tablets x 3 daily
  Arms: Placebo (Hydralazine Isosorbide Dinitrate)
Drug: Metformin Hydrochloride — Tablet Metformin hydrochloride 500 mg 2 tablets x 2 daily (eGFR 35-60 ml/min: 500 mg x 2 daily)
  Arms: Metformin
Drug: Placebo Oral Tablet — 2 tablets x 2 daily (eGFR 35-60 ml/min: 500 mg x 2 daily)
  Arms: Placebo (Metformin)

SUMMARY:
The present study is testing in a combined design to types of drugs in patients with chronic heart failure: 1) Hydralazine in combination with isosorbide dinitrate (BiDil) and 2) Metformin hydrochloride. The study is double blind, placebo controlled.

1. The first hypothesis is that hydralazine in combination with isosorbide dinitrate can reduce mortality and hospitalization with worsening heart failure in chronic heart failure patients with reduced LVEF.
2. The second hypothesis is that treatment with metformin in chronic heart failure patients with reduced LVEF and type 2 diabetes / diabetes risk / insulin resistance can reduce mortality and cardiovascular hospitalizations. Among secondary endpoints are reduction in new-onset diabetes in heart failure patients with insulin resistance and diabetes risk profile and patient safety.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria for both H-HeFT and Met-HeFT

* Patients with chronic heart failure
* NYHA-class II, III or IV
* LVEF </= 40% within 12 months prior to screening. The echocardiography should (i) be performed after uptitration in heart failure medication and (ii) LVEF from the most recently performed echocardiographic study should be used and (iii) LVEF must not be measured during rapid atrial fibrillation, i.e. heart rate >110/min) and (iiii) the echocardiography should be performed at least 3 months after CRT-implantation.
* Patients should be uptitrated to recommended or maximally tolerated dose of ACE-I/ARB/ARNI (unless contraindicated) and beta-blocker (unless contraindicated). If indicated, an aldosterone receptor antagonist should be given (unless contraindicated).
* A CRT device should be implanted, if indicated and accepted by the patient and patients with a CRT device should be treated for > 3 months.
* Implantation of an ICD unit should be planned or already done, if indicated and accepted by the patient. The patient can be included in the study before a planned ICD implantation has been performed.
* Informed consent

Specific inclusion criteria for only H-HeFT:

* Systolic blood pressure ≥100 mmHg
* NT-proBNP > 350 pg/ml or BNP > 80 pg/ml (in patients treated with ARNI, NT-proBNP must be used)

Specific inclusion criteria for only Met-HeFT:

Patients must have a diagnosis of type 2 diabetes or insulin resistance or diabetes risk. This includes 1 or more of any of the following:

* A previous diagnosis of type 2 diabetes at any time without Metformin treatment during the last 3 months
* HbA1c ≥ 5.5 % (≥ 37 mmol/mol) within 12 months prior to screening
* Fasting P-glucose ≥ 5.6 mmol/l within 12 months prior to screening (measured when the patient in stable condition / has no intercurrent illness)
* Body mass index ≥ 30 kg/m2
* If oral glucose tolerance testing (OGTT) has been performed at any time prior to randomization: 2 hour P-glucose ≥ 7.8 mmol/l
* In addition, patients in Met-HeFT must have eGFR ≥ 35 ml/min (MDRD)

Patients are randomized through an internet based randomization module. Patients can be allocated to a) both H-HeFT and Met-HeFT or to b) only H-HeFT or to c) only Met-HeFT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
H-HeFT combined primary endpoint | Through study completion, an average of 4 years
  Combined endpoint: Death or hospitalization with worsening heart failure or an urgent visit resulting in intravenous therapy or metolazone therapy for heart failure or heart transplantation or implantation of a LVAD.
Met-HeFT combined primary endpoint | Through study completion, an average of 4 years
  Combined endpoint: Death or hospitalization with worsening heart failure or an urgent visit resulting in intravenous therapy or metolazone therapy for heart failure or heart transplantation or implantation of a LVAD or acute myocardial infarction or stroke

SECONDARY OUTCOMES:
H-HeFT Death | Through study completion, an average of 4 years
  Death
H-HeFT: Heart failure events | Through study completion, an average of 4 years
  Hospitalization with worsening heart failure or urgent visit resulting in intravenous therapy or metolazone therapy for heart failure or heart transplantation or implantation of LVAD
H-HeFT: Death or cardiovascular hospitalization | Through study completion, an average of 4 years
  Combined endpoint: Death or cardiovascular hospitalizations (hospitalization with worsening heart failure, acute myocardial infarction, or stroke) or urgent visit resulting in intravenous therapy or metolazone therapy for heart failure or or heart transplantation or implantation of LVAD
H-HeFT combined primary endpoint of total (first and recurrent) events | Through study completion, an average of 4 years
  Composite of total (first and recurrent) events in the primary endpoint:
  Death or hospitalization with worsening heart failure or an urgent visit resulting in intravenous therapy or metolazone therapy for heart failure or heart transplantation or implantation of a LVAD.
H-HeFT: All-cause, total (first and subsequent) hospitalizations | Through study completion, an average of 4 years
  Any hospitalization
H-HeFT: Change in NT-proBNP from baseline to final follow-up | Through study completion, an average of 4 years
  Change in NT-proBNP from baseline to final follow-up
H-HeFT: Cardiovascular hospitalizations | Through study completion, an average of 4 years
  Any cardiovascular hospitalization
Met-HeFT combined endpoint of total (first and recurrent) events in the primary endpoint | Through study completion, an average of 4 years
  Combined endpoint of total (first and recurrent) events: Death or hospitalization with worsening heart failure or an urgent visit resulting in intravenous therapy or metolazone therapy for heart failure or heart transplantation or implantation of a LVAD or acute myocardial infarction or stroke
Met-HeFT secondary endpoint: Death | Through study completion, an average of 4 years
  Death
Met-HeFT: Hospitalization with worsening heart failure or urgent visit resulting in intravenous therapy or metolazone therapy for heart failure or heart transplantation or implantation of a LVAD | Through study completion, an average of 4 years
  Hospitalization with worsening heart failure or urgent visit resulting in intravenous therapy or metolazone therapy for heart failure or heart transplantation or implantation of a LVAD
Met-HeFT Extended clinical endpoint (first event analysis): The primary endpoint or coronary revascularization or non-coronary revascularization or limb amputation. | Through study completion, an average of 4 years
  Met-HeFT: Extended clinical endpoint (first event analysis): The primary endpoint or coronary revascularization or non-coronary revascularization or limb amputation.
Met-HeFT secondary endpoint: Acute myocardial infarction | Through study completion, an average of 4 years
  Acute myocardial infarction
Met-HeFT secondary endpoint: Stroke | Through study completion, an average of 4 years
  Stroke
Met-HeFT secondary endpoint: New onset type 2 diabetes | Through study completion, an average of 4 years
  New onset type 2 diabetes
Met-HeFT secondary endpoint: Hospitalization or death caused by lactic acidosis. | Through study completion, an average of 4 years
  Hospitalization or death caused by lactic acidosis.
Met-HeFT: All-cause, total (first and subsequent) hospitalizations | Through study completion, an average of 4 years
  Any hospitalization
Met-HeFT: Change in NT-proBNP from baseline to final follow-up | Through study completion, an average of 4 years
  Change in NT-proBNP
Met-HeFT: Cardiovascular hospitalizations | Through study completion, an average of 4 years
  Any cardiovascular hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Wiggers, MD, PhD, Study Chair — Dept. of Cardiology, Aarhus University Hospital, Aarhus, Denmark; Lars Køber, MD, PhD, Study Chair — Dept. of Cardiology, Rigshospitalet, Copenhagen, Denmark; Finn Gustafsson, MD, PhD, Principal Investigator — Dept. of Cardiology, Rigshospitalet, Copenhagen, Denmark; Søren Mellemkjaer, MD, PhD, Principal Investigator — Dept. of Cardiology, Aarhus University Hospital, Aarhus, Denmark; Gunnar Gislason, MD, PhD, Study Chair — The Danish Heart Foundation, Copenhagen, Denmark
Locations (26):
- Denmark (26):
  - Holbæk Hospital, Holbæk, Region Sjælland
  - Sygehus Sønderjylland, Aabenraa, Aabenraa
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Amager Hospital, Copenhagen
  - Bispebjerg Hospital, Copenhagen
  - Gentofte Hospital, Copenhagen
  - Glostrup Hospital, Copenhagen
  - Herlev Hospital, Copenhagen
  - Hvidovre Hospital, Copenhagen
  - Rigshospitalet, Copenhagen
  - Sydvestjysk Sygehus, Esbjerg, Esbjerg
  - Herning Hospital, Herning
  - Nordsjællands Hospital Hillerød, Hillerød
  - Regionshospital Nordjylland, Hjørring, Hjørring
  - Holbæk Hospital, Holbæk
  - Horsens Hospital, Horsens
  - Kolding Hospital, Kolding
  - Nykøbing Falster Hospital, Nykøbing Falster
  - Odense University Hospital, Odense
  - Randers Hospital, Randers
  - Sjællands Universitetshospital, Roskilde, Roskilde
  - Silkeborg Hospital, Silkeborg
  - Slagelse Sygehus, Slagelse
  - Vejle Hospital, Vejle
  - Viborg Hospital, Viborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wiggers H, Kober L, Gislason G, Schou M, Poulsen MK, Vraa S, Nielsen OW, Bruun NE, Norrelund H, Hollingdal M, Barasa A, Bottcher M, Dodt K, Hansen VB, Nielsen G, Knudsen AS, Lomholdt J, Mikkelsen KV, Jonczy B, Bronnum-Schou J, Poenaru MP, Abdulla J, Raymond I, Mahboubi K, Sillesen K, Serup-Hansen K, Madsen JS, Kristensen SL, Larsen AH, Botker HE, Torp-Petersen C, Eiskjaer H, Moller J, Hassager C, Steffensen FH, Bibby BM, Refsgaard J, Hofsten DE, Mellemkjaer S, Gustafsson F. The DANish randomized, double-blind, placebo controlled trial in patients with chronic HEART failure (DANHEART): A 2 x 2 factorial trial of hydralazine-isosorbide dinitrate in patients with chronic heart failure (H-HeFT) and metformin in patients with chronic heart failure and diabetes or prediabetes (Met-HeFT). Am Heart J. 2021 Jan;231:137-146. doi: 10.1016/j.ahj.2020.09.020. Epub 2020 Oct 9. PMID 33039340